CLINICAL TRIAL: NCT01027000
Title: Phase II Study of Reduced-Intensity Allogeneic Stem Cell Transplant for High-Risk Chronic Lymphocytic Leukemia (CLL)
Brief Title: Donor Stem Cell Transplant in Treating Patients With High-Risk Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Genentech, Inc. (Industry); Biologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB 100701; CDR0000660555 (Registry Identifier: Physician Data Query); U10CA031946 (NIH); NCI-2011-01995 (Registry Identifier: NCI Clinical Trials Reporting Office)
Record Dates: First submitted 2009-12-04; First posted 2009-12-07 (Estimated); Results first posted 2017-05-03 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Leukemia; Lymphoma
Keywords: refractory chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; B-cell chronic lymphocytic leukemia; contiguous stage II small lymphocytic lymphoma; noncontiguous stage II small lymphocytic lymphoma; recurrent small lymphocytic lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; Busulfan; Cyclophosphamide; fludarabine phosphate; Methotrexate; Sirolimus; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Combination of chemotherapy and transplant) (Experimental): See detailed description
  Interventions: Biological: rituximab; Drug: busulfan; Drug: cyclophosphamide; Drug: fludarabine phosphate; Drug: methotrexate; Drug: sirolimus; Drug: tacrolimus; Procedure: allogeneic stem cell transplant

INTERVENTIONS:
Biological: rituximab
Drug: busulfan
Drug: cyclophosphamide
Drug: fludarabine phosphate
Drug: methotrexate
Drug: sirolimus
Drug: tacrolimus
Procedure: allogeneic stem cell transplant

SUMMARY:
RATIONALE: Giving low doses of chemotherapy before a donor stem cell transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. Also, monoclonal antibodies, such as rituximab, can find cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving tacrolimus, sirolimus, and methotrexate after the transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well donor stem cell transplant works in treating patients with high-risk chronic lymphocytic leukemia or small lymphocytic lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if this treatment can improve 2-year current progression-free survival (PFS) in the early disease cohort compared to historical controls. Specifically, we plan to study whether we can achieve 2-year PFS ≥ 70% and to exclude 2 year PFS ≤ 50%

Secondary

* To determine whether in the advanced disease cohort we can achieve 2-year current PFS ≥ 50% and to exclude 2-year PFS ≤ 30%
* To assess objective response rate.
* To assess the incidence of grade 2-4 and 3-4 acute graft-vs-host disease (GVHD).
* To assess the incidence of extensive chronic GVHD.
* To assess the incidence of treatment-related mortality at 100 days and 1 year
* To assess overall survival
* To assess donor chimerism for CD3+ cells at 1 and 2 years after transplantation
* To investigate the presence of donor antigen-specific T-cell clones before and after withdrawal of immune suppression.
* To compare the relapse profiles of patients with T-cell responses against CLL to those whose CLL cells are not reactive
* To prospectively examine the impact of high-risk genomic features and immune-based single nucleotide polymorphisms on response, toxicity, and 2-year PFS to reduced intensity allogeneic stem cell transplant

OUTLINE: This is a multicenter study.

* Preparative regimen: Patients receive 1 of 2 preparative regimens at the discretion of the participating institution.

  * Preparative regimen 1: Patients receive rituximab IV on days -7, -1, 7, and 14 and fludarabine phosphate IV over 30 minutes and busulfan IV over 3 hours on days -5 to -2. .
  * Preparative regimen 2: Patients receive rituximab IV on days -7, -1, 7, and 14, fludarabine phosphate IV over 30 minutes on days -5 to -2, and cyclophosphamide IV over 1-2 hours on days -5 to -3. Patients with matched unrelated donors also receive anti-thymocyte globulin IV over 4-6 hours on days -6 to -4.
* Graft-vs-host disease (GVHD) prophylaxis: Patients who receive preparative regimen 1 may receive either GVHD prophylaxis regimen 1 or 2; patients who receive preparative regimen 2 may only receive GVHD prophylaxis regimen 2.

  * GVHD prophylaxis regimen 1: Patients receive tacrolimus either orally or IV and oral sirolimus beginning on day -2 and continuing until day 60, followed by a taper until day 180. Patients also receive methotrexate IV on days 1, 3, and 6.
  * GVHD prophylaxis regimen 2: Patients receive tacrolimus either orally or IV beginning on day -2 and continuing until day 60, followed by a taper until day 180. Patients also receive methotrexate IV on days 1, 3, 6, and 11.
* Transplantation: Patients undergo allogeneic peripheral blood stem cell transplantation on day 0.
* Maintenance therapy: Patients receive rituximab IV at 3, 6, 9, and 12 months after transplantation.

Peripheral blood and bone marrow aspirate samples may be collected periodically for correlative laboratory studies.

Patients are followed up periodically for a maximum of 5 years from study entry.

ELIGIBILITY:
Patient Eligibility:

1. Diagnosis of B-cell chronic lymphocytic leukemia or B-cell small lymphocytic lymphoma.

   Diagnosis should be according to International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2008 Criteria
   1. Early Disease Cohort - Patients in the early disease cohort must include one or more of the following:

      * FISH showing deletion 17p in ≥ 20% of cells (either at diagnosis or any time prior to study entry) either alone or in combination with other cytogenetic abnormalities
      * FISH showing del 11q in ≥ 20% of cells (either at diagnosis or any time prior to study entry) either alone or in combination with other cytogenetic abnormalities, unless the patient has achieved a complete remission by IWCLL 2008 which includes CT scan, bone marrow morphology and flow cytometry
      * Failure to achieve a partial response with initial chemotherapy, but with lack of progression. These patients may receive a second therapy to improve their response prior to transplant.
      * Patients who, at the time of first progression, have a 17p deletion by FISH in ≥ 20% of cells, either alone or in combination with other cytogenetic abnormalities.

      The duration of the first progression is not specified.
      * In addition, patients in the early disease cohort must have all of the following:

        * Received at least 2 cycles of induction therapy. It is expected that most patients will receive at least 4 months of therapy prior to enrollment, but this is not required. Suggested regimens include but are not limited to the following: fludarabine plus rituximab, fludarabine, cyclophosphamide plus rituximab, pentostatin, cyclophosphamide plus rituximab, bendumustine plus rituximab, or alemtuzumab alone or in combination with other agents. Patients may receive no more than 2 different regimens prior to proceeding to transplantation.
        * Nodes ≤ 5 cm
   2. Advanced Disease Cohort - Patients in the advanced disease cohort must include one or more of the following:

      * FISH showing deletion 17p in ≥ 20% of cells (regardless of interval from initial therapy) either alone or in combination with other cytogenetic abnormalities
      * First progression < 24 months after completing therapy. This includes progression on initial therapy.
      * Second or subsequent progression
      * In addition, patients in the advanced disease cohort must have all of the following:

        * Stable disease or better by the Revised IWCLL 2008 NCI Criteria to their most recent chemotherapy
        * Nodes ≤ 5 cm
2. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
3. Age Requirement - Patients must be between ≥ 18 and < 70 years of age
4. Cytotoxic Chemotherapy or Alemtuzamab - There must be at least 4 weeks after day 1 of the last cycle of cytotoxic chemotherapy, or alemtuzamab.
5. Human Immunodeficiency Virus (HIV) Status - Patients must have no HIV infection.

   Allogeneic transplantation in the HIV patient population is not well-defined and there are likely to be requirements for concomitant anti-HIV therapy and anti-GVHD therapy that would create potentially dangerous pharmacokinetic interactions among the different agents that could constrain therapeutic options for controlling both HIV and GVHD.
6. Hepatitis B and C - Patients must have no Hepatitis B sAg, anti-HBc or HCV.
7. Diffusion capacity of carbon monoxide DLCO must be ≥ 40% predicted
8. Left ventricular ejection fraction (LVEF) by Echocardiogram (ECHO) or Multiple gated acquisition (MUGA) must be ≥ 30%
9. Diabetes or Serious Infection - Patients must have no uncontrolled diabetes mellitus or active uncontrolled serious infections
10. Pregnancy and Nursing Status - Patients must be non-pregnant and non-nursing. Treatment under this protocol would expose a fetus to significant risks. Women of childbearing potential should have a negative pregnancy test prior to study entry.

    Women and men of reproductive potential should agree to use an appropriate method of birth control throughout their participation in this study due to the teratogenic potential of the therapy utilized in this trial. Appropriate methods of birth control include oral contraceptives, implantable hormonal contraceptives (Norplant®), or double barrier method (diaphragm plus condom).
11. Richter's Transformation - Patients must have no history of Richter's transformation.
12. Initial Required Laboratory Values:

    * Serum Creatinine < 2 mg/dL
    * Calculated Creatinine Clearance ≥ 40 mL/min
    * AST < 3 x ULN
    * Total Bilirubin < 2 mg/dL (except for Gilbert's syndrome)

Donor Eligibility:

1. Donors may be either a 6/6 HLA-matched related donor by low-resolution typing at HLA A, B, DR.
2. Donors may be an 8/8 HLA-matched unrelated donor at HLA A, B, C, DR. Unrelated donors will be analyzed by molecular typing at both HLA Class I and Class II (A, B, C, DR loci).
3. Syngeneic donors are not eligible
4. Donors must be healthy and must be an acceptable donor as per institutional standards for stem cell donation.
5. There will be no donor age restriction.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2010-02; Primary Completion 2016-01 (Actual); Study Completion 2023-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edwin P. Alyea, MD, Study Chair — Dana-Farber Cancer Institute
Locations (25):
- United States (25):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Union Hospital of Cecil County, Elkton, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Monter Cancer Center of the North Shore-LIJ Health System, Lake Success, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between February 2010 and January 2014, 68 participants were recruited.
Groups:
- Treatment (Combination of Chemotherapy and Transplant): Preparative: Patients receive 1 of 2 preparative regimens (Reg) chosen by the treating institution
  * Reg1: Rituximab (RTX) 500 mg/m^2 IV on days -7, -1, 7, and 14 & fludarabine phosphate (FP) 30 mg/m^2 IV & busulfan 0.8 mg/kg IV on days -5 to -2
  * Reg 2: RTX 500 mg/m^2 IV on days -7, -1, 7, and 14 & FP 30 mg/m^2 IV on days -5 to -2 & cyclophosphamide 1 g/m^2 IV on days -5 to -3
  Graft-vs-host disease (GVHD) prophylaxis: Patients treated with preparative regimen 1 received either GVHD prophylaxis regimen 1 or 2; those given preparative regimen 2 received regimen 2
  * Reg 1: Tacrolimus PO or IV & oral sirolimus 12 mg on day -2 through day 60, followed by taper until day 180 & methotrexate (MTX) 5 mg/m^2 IV on days 1, 3, and 6.
  * Reg 2: Tacrolimus PO or IV on day -2 through day 60, followed by taper until day 180 & MTX 5mg/m^2 IV on days 1, 3, 6, & 11 Transplantation: allogeneic peripheral blood transplant on day 0 Maintenance: RTX 500 mg/m^2 IV at 3, 6, 9, & 12 months post-transplant
Period: Overall Study
Arm/Group | Treatment (Combination of Chemotherapy and Transplant)
Started | 68
Completed | 68
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Combination of Chemotherapy and Transplant)
Number analyzed (Participants) | 68
Age, Continuous [Median (Full Range); unit: years] | 56 [26 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 62
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 66
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 68
Disease stage [Number; unit: participants] — Early Disease: Participants must have received ≥2 cycles of induction therapy & have nodes ≤ 5 cm with one or more of the following: FISH deletion 17p, FISH del 11q, failure to achieve a partial response with initial chemotherapy with no progression, or have a 17p deletion by FISH at the time of first progression
  Advanced Disease: Participants must have stable disease or better to their most recent chemotherapy & have nodes ≤ 5 cm with one or more of the following:
  FISH deletion 17p, first progression < 24 months after completing therapy, or a subsequent progression
  participants
    Early Disease | 14
    Advanced Disease | 50
    Not reported | 4

OUTCOME MEASURES:

1. Primary Outcome: 2-year Progression-free Survival in Early Disease Participants
Description: Percentage of participants who were alive and progression free at 2 years for participants with early disease stage. The 2 year progression free survival, with 95% confidence interval, was estimated using the Kaplan Meier method.
  A progression is defined as one of the following events:
  * >= 50% increase in the products of at least two lymph nodes on two consecutive determinations two weeks apart (at least one lymph node must be >= 2 cm); appearance of new palpable lymph nodes.
  * >= 50% increase in the size of the liver and/or spleen as determined by measurement below the respective costal margin; appearance of palpable hepatomegaly or splenomegaly, which was not previously present.
  * > 50% increase in peripheral blood lymphocytes with an absolute increase > 5000/μL.
  * Transformation to a more aggressive histology (i.e., Richter's syndrome or prolymphocytic leukemia with >= 56% prolymphocytes).
Time Frame: 2 years post-registration
Population: Participants with early disease stage were analyzed. Two participants, who did not start protocol therapy, were excluded from this analysis.
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Combination of Chemotherapy and Transplant)
Number analyzed (Participants) | 12
percentage of participants | 79.5 [39 to 94.5]

2. Secondary Outcome: Response
Time Frame: 5 years post-registration
Reporting Status: Not Posted

3. Secondary Outcome: Acute Graft-vs-host Disease (GVHD)
Time Frame: 5 years post-registration
Reporting Status: Not Posted

4. Secondary Outcome: Chronic GVHD
Time Frame: 5 years post-registration
Reporting Status: Not Posted

5. Secondary Outcome: Treatment-related Mortality
Time Frame: 6 months post-transplant
Reporting Status: Not Posted

6. Secondary Outcome: Overall Survival
Time Frame: 5 years post-registration
Reporting Status: Not Posted

7. Secondary Outcome: Chimerism for CD3
Time Frame: 5 years post-registration
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Adverse event data is available for 59 participants . The remaining 9 participants cancelled before beginning treatment or withdrew consent for follow-up.
Arm/Group | Treatment (Combination of Chemotherapy and Transplant)
Serious Adverse Events (participants affected / at risk) | 6/59
Other Adverse Events (participants affected / at risk) | 58/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Combination of Chemotherapy and Transplant) (N=59)
Anemia (Blood and lymphatic system disorders) | 5 (8)
Vertigo (Ear and labyrinth disorders) | 1 (3)
Corneal ulcer (Eye disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1)
Keratitis (Eye disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (3)
Vomiting (Gastrointestinal disorders) | 1 (3)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Vaginal infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2)
Cholesterol high (Investigations) | 1 (1)
Creatinine increased (Investigations) | 4 (5)
Investigations - Other, specify (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (5)
Neutrophil count decreased (Investigations) | 4 (6)
Platelet count decreased (Investigations) | 6 (7)
White blood cell decreased (Investigations) | 3 (4)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (6)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (3)
Dysphasia (Nervous system disorders) | 1 (1)
Edema cerebral (Nervous system disorders) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 2 (2)
Nervous system disorders - Other, specify (Nervous system disorders) | 2 (4)
Stroke (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Genital edema (Reproductive system and breast disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4)
Hypertension (Vascular disorders) | 3 (3)
Hypotension (Vascular disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Combination of Chemotherapy and Transplant) (N=59)
Anemia (Blood and lymphatic system disorders) | 48 (161)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 (7)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 5 (5)
Atrioventricular block first degree (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Restrictive cardiomyopathy (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 4 (5)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (4)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Cushingoid (Endocrine disorders) | 3 (4)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (4)
Blurred vision (Eye disorders) | 3 (3)
Cataract (Eye disorders) | 1 (1)
Corneal ulcer (Eye disorders) | 1 (2)
Dry eye (Eye disorders) | 6 (11)
Eye disorders - Other, specify (Eye disorders) | 5 (7)
Eye pain (Eye disorders) | 1 (1)
Keratitis (Eye disorders) | 1 (1)
Papilledema (Eye disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Scleral disorder (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 4 (7)
Abdominal pain (Gastrointestinal disorders) | 13 (21)
Ascites (Gastrointestinal disorders) | 2 (6)
Colonic ulcer (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 11 (14)
Diarrhea (Gastrointestinal disorders) | 28 (54)
Dry mouth (Gastrointestinal disorders) | 6 (16)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 3 (3)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 4 (4)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (3)
Hemorrhoids (Gastrointestinal disorders) | 2 (2)
Ileus (Gastrointestinal disorders) | 1 (1)
Lip pain (Gastrointestinal disorders) | 1 (1)
Malabsorption (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 9 (9)
Nausea (Gastrointestinal disorders) | 29 (64)
Oral pain (Gastrointestinal disorders) | 3 (4)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 2 (2)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 17 (28)
Chills (General disorders) | 8 (11)
Edema face (General disorders) | 5 (5)
Edema limbs (General disorders) | 17 (42)
Fatigue (General disorders) | 34 (105)
Fever (General disorders) | 17 (22)
Infusion related reaction (General disorders) | 2 (2)
Injection site reaction (General disorders) | 1 (1)
Irritability (General disorders) | 2 (2)
Localized edema (General disorders) | 1 (1)
Malaise (General disorders) | 3 (3)
Neck edema (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2)
Pain (General disorders) | 4 (8)
Cholecystitis (Hepatobiliary disorders) | 2 (3)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 5 (10)
Allergic reaction (Immune system disorders) | 2 (2)
Abdominal infection (Infections and infestations) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 2 (2)
Eye infection (Infections and infestations) | 1 (1)
Hepatic infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 9 (14)
Joint infection (Infections and infestations) | 1 (1)
Lip infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 8 (9)
Meningitis (Infections and infestations) | 1 (1)
Mucosal infection (Infections and infestations) | 2 (4)
Rhinitis infective (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 2 (9)
Skin infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 9 (15)
Urinary tract infection (Infections and infestations) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (3)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Intraoperative renal injury (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 7 (8)
Alanine aminotransferase increased (Investigations) | 26 (65)
Alkaline phosphatase increased (Investigations) | 17 (37)
Aspartate aminotransferase increased (Investigations) | 25 (71)
Blood bilirubin increased (Investigations) | 21 (44)
Cholesterol high (Investigations) | 8 (12)
Creatinine increased (Investigations) | 36 (70)
INR increased (Investigations) | 1 (1)
Investigations - Other, specify (Investigations) | 13 (51)
Lymphocyte count decreased (Investigations) | 35 (97)
Lymphocyte count increased (Investigations) | 7 (9)
Neutrophil count decreased (Investigations) | 51 (137)
Platelet count decreased (Investigations) | 52 (143)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 7 (9)
White blood cell decreased (Investigations) | 33 (80)
Anorexia (Metabolism and nutrition disorders) | 10 (14)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 40 (153)
Hyperkalemia (Metabolism and nutrition disorders) | 14 (22)
Hypermagnesemia (Metabolism and nutrition disorders) | 4 (4)
Hypernatremia (Metabolism and nutrition disorders) | 7 (9)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 14 (19)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 19 (34)
Hypocalcemia (Metabolism and nutrition disorders) | 26 (50)
Hypoglycemia (Metabolism and nutrition disorders) | 4 (5)
Hypokalemia (Metabolism and nutrition disorders) | 13 (18)
Hypomagnesemia (Metabolism and nutrition disorders) | 25 (52)
Hyponatremia (Metabolism and nutrition disorders) | 18 (39)
Hypophosphatemia (Metabolism and nutrition disorders) | 12 (22)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 4 (9)
Obesity (Metabolism and nutrition disorders) | 9 (27)
Abdominal soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (12)
Arthritis (Musculoskeletal and connective tissue disorders) | 4 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (21)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (6)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 4 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (9)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (5)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3)
Ataxia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 7 (11)
Dysesthesia (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 3 (4)
Headache (Nervous system disorders) | 23 (31)
Lethargy (Nervous system disorders) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 2 (3)
Paresthesia (Nervous system disorders) | 2 (3)
Peripheral motor neuropathy (Nervous system disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (14)
Sinus pain (Nervous system disorders) | 3 (5)
Stroke (Nervous system disorders) | 1 (2)
Syncope (Nervous system disorders) | 1 (1)
Transient ischemic attacks (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 14 (25)
Agitation (Psychiatric disorders) | 1 (4)
Anxiety (Psychiatric disorders) | 7 (16)
Confusion (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 7 (12)
Hallucinations (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 8 (9)
Libido decreased (Psychiatric disorders) | 2 (2)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Cystitis noninfective (Renal and urinary disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 2 (3)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 3 (6)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 1 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (9)
Apnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 22 (44)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15 (28)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 5 (10)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (12)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Periorbital edema (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (20)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 33 (68)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 10 (12)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 4 (5)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (2)
Flushing (Vascular disorders) | 2 (2)
Hot flashes (Vascular disorders) | 2 (4)
Hypertension (Vascular disorders) | 25 (76)
Hypotension (Vascular disorders) | 5 (5)
Superficial thrombophlebitis (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less